CLINICAL TRIAL: NCT01926405
Title: Evaluation of Excessive Diurnal Sleepiness by the Expression and Activity of Salivary Amylase in Children With Hypersomnia.
Brief Title: Amylase and Hypersomnia
Acronym: Amylase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011.681
Record Dates: First submitted 2013-08-12; First posted 2013-08-20 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Hypersomnia in Children
Keywords: hypersomnia; narcolepsy; amylase; salivary sampling
MeSH Terms: conditions — Disorders of Excessive Somnolence; Narcolepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects with narcolepsy or with idiopathic hypersomnia (Other)
  Interventions: Procedure: saliva collection
- Control patients with no sleeping disorder (Other)
  Interventions: Procedure: saliva collection

INTERVENTIONS:
Procedure: saliva collection — collection of saliva

SUMMARY:
Hypersomnia is defined as a reduced ability to remain awake during the day. There are basically two types of central hypersomnia: narcolepsy and idiopathic hypersomnia. Currently, the diagnosis of these sleep disorders is based on polysomnographic recordings which is difficult to access. Tests of sleepiness (Epworth, Karolinska) are subjective.

A biological marker of sleepiness, easily accessible and measurable, would be very useful for the diagnosis and therapeutic follow up of excessive diurnal sleepiness. Salivary secretions appear as good physiological markers. Studies have shown for healthy subjects, that the expression and activity of salivary amylase are increased when subjects are deprived of sleep.

The investigators propose to explore the usefulness of salivary biomarkers (including amylase) as a new non-invasive and simple technique for the assessment of excessive daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

Subjects with hypersomnia (narcolepsy or idiopathic):

* Children and adolescents with hypersomnia (according to ICSD diagnostic criteria 2); narcolepsy or idiopathic hypersomnia (with or without lengthening of sleep),
* aged > 6 years and <18 years,
* no treatment,
* Parent consent

Control subjects:

* healthy children and adolescents without any known pathology,
* aged > 6 years and <18 years,
* matched on sex and age> 6 years - <12 years,> 12 - <18 years)
* Parent Consent

Exclusion Criteria:

* Subjects with hypersomnia (narcolepsy or idiopathic):
* Secondary narcolepsy,
* Symptomatic hypersomnia,
* Restless legs syndrome,
* Sleep apnea syndrome,
* Severe neurological, psychiatric, cognitive or endocrinological concomitant disease.

Control subjects:

* Hypersomnia,
* Restless legs syndrome,
* Sleep apnea syndrome,
* Severe neurological, psychiatric, cognitive or endocrinological concomitant disease,
* Sleep disorder evaluated by a score > 70 on the Sleep Disturbance Scale for Children19,
* Excessive daytime sleepiness according to Epworth scales (score > 10),
* Abnormal sleep time according to the age (sleep diary).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Determination of the expression and enzymatic activity of salivary amylase. | 3 days
  Show an increase of salivary amylase for children with hypersomnia or narcolepsy compared to a group of children matched on age and sex.

SECONDARY OUTCOMES:
Measurement of the mean sleep onset latency using the Multiple Sleep Latency Test (MSLT) | 3 days
  To highlight a correlation between the degree of somnolence measured by MSLT and the rate of salivary amylase.
Measurement of the somnolence using Epworth and Karolinska scales | 3 days
  To highlight a correlation between the degree of somnolence measured by the scales and the rate of salivary amylase.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant, Exploration et pathologie du sommeil, Bron, France